CLINICAL TRIAL: NCT03472651
Title: Interventional, Randomized, Single Dose, Open-label, Crossover, Bioequivalence Study in Healthy Men and Women to Compare Two Pharmaceutical Formulations of Flupentixol/Melitracen (Deanxit®) - in Fasted and Fed Conditions
Brief Title: Bioequivalence Study to Compare Two Formulations of Deanxit®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17686A
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — flupentixol, melitracen drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A1 Fasted condition (Experimental): Subjects in cohort A1 will be administered the Investigational Medicinal Product in a fasted state, 30 subjects per cohort
  Interventions: Drug: test treatment: flupentixol/melitracen; Drug: reference treatment: flupentixol/melitracen
- Cohort A2 Fed condition (Experimental): Subjects in cohort A2 will be administered the Investigational Medicinal Product in a fed state, 30 subjects per cohort
  Interventions: Drug: test treatment: flupentixol/melitracen; Drug: reference treatment: flupentixol/melitracen

INTERVENTIONS:
Drug: test treatment: flupentixol/melitracen — 0.5 mg flupentixol and 10 mg melitracen, film-coated tablet, single dose
Drug: reference treatment: flupentixol/melitracen — 0.5 mg flupentixol and 10 mg melitracen, coated tablet, single dose
  Other Names: Deanxit®

SUMMARY:
The purpose of this study is to establish bioequivalence of flupentixol/meltracen, between a new film-coated tablet formulation and the marketed coated tablet formulation (Deanxit®), administered single dose in fasted and fed condition

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥18 and ≤55 years of age with a body mass index (BMI) of ≥ 18.5 and ≤ 28 kg/m2.
* Women must be non-pregnant and non-lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
AUC0-72h: flupentixol | from zero to 72 hours post-dose
  the area under the flupentixol plasma concentration-time curve
Cmax: flupentixol | from zero to 72 hours post-dose
  maximum observed plasma concentration of flupentixol
AUC0-72h: melitracen | from zero to 72 hours post-dose
  the area under the melitracen plasma concentration-time curve
Cmax: melitracen | from zero to 72 hours post-dose
  maximum observed concentration of melitracen

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- CN1036 Shijitan Hospital, Beijing, China